CLINICAL TRIAL: NCT03721731
Title: A Post-Market Surveillance Study Examining the Safety & Effectiveness of Using the g-Cath EZ Delivery Catheter With Snowshoe Suture Anchors and Associated Devices (g-Prox EZ, g-Lix and Transport) for the Treatment of Obesity
Brief Title: A Post-Market Surveillance Study of Using the g-Cath EZ for Treating Obesity
Status: Completed | Type: Observational
Sponsor: USGI Medical (Industry)
Collaborators: Centro Medico Teknon (Other); Hospital Universitario Madrid Sanchinarro (Other)
Responsible Party: Sponsor
Other Study IDs: 50518 TPR
Record Dates: First submitted 2018-10-22; First posted 2018-10-26 (Actual); Last update posted 2020-11-04 (Actual); Status verified 2018-10

CONDITIONS: Treatment of Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

INTERVENTIONS:
Device: Obesity treatment with a Plication device — Plicating the stomach to treat obesity

SUMMARY:
This is a multi-center, prospective study evaluating a treatment for obesity.

DETAILED DESCRIPTION:
This is a multi-center, prospective study evaluating a treatment for obesity using the g-Cath EZ and associated devices. The intent is to evaluate the safety and efficacy of a modified Snowshoe suture anchor placement pattern called Pose 2 (suture anchors placed in the mid + distal body of the stomach, with none placed in the fundus) along with a moderate intensity diet and exercise program. The g-Cath EZ and the associated devices (the g-Prox EZ, g-Lix & Transport) are known collectively as the Incisionless Operating Platform (IOP). Efficacy of the treatment will be evaluated based on changes in weight loss over 12 months, & adverse events will be recorded throughout the duration of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form
2. Subject agrees to be compliant with study requirements and adhere to post-operative dietary & exercise recommendations for the duration of the study.
3. Subjects between the ages of 22-60 years.
4. If female, be either post-menopausal, surgically sterile or agree to practice birth control during year of study and have negative serum HCG at screening/baseline.
5. Have a Body Mass Index (BMI) of ≥ 35 and < 40 with one obesity related co-morbid condition (defined by 1991 NIH Guidelines with document referenced by FDA (Appropriateness Criteria for Bariatric Surgery: Beyond the NIH Guidelines)).

   1. Pre-diabetes - Fasting plasma glucose test >100 mg/dl but ≤125 or oral glucose tolerance test ≥140 mg/dl but <200.
   2. Diabetes - Individuals taking insulin and/or oral hypoglycemic medications or have a fasting glucose >126 mg/dl.
   3. Hypertension - SBP>140 or DBP>90 or the use of an antihypertensive medication
   4. Dyslipidemia - Triglycerides > 250 mg/dl or cholesterol > 220 mg/dl or HDL < 35 mg/dl or LDL > 200 or use of lipid lowering medications.
   5. Sleep Apnea - A formal sleep study test consistent with this diagnosis; Epworth sleepiness scale ≥ 6; Polysomnography with respiratory disturbance index ≥ 10 hyponeic and/or apneic episodes per hour of sleep.
   6. Venous Stasis Disease - Presence or history of pretibial venous stasis ulcers.
   7. Chronic Joint Disease - Deterioration of joint cartilage and the formation of new bone (bone spurs) at the margins of the joints.
   8. Quality of Life - Impaired quality of life is defined as poor quality of life as measured by a formal and previously validated quality of life (QOL) questionnaire (e.g. SF-12)
   9. Gastroesophageal Reflux - Heartburn regurgitation or pain with swallowing and chest pain. Symptoms relieved by antacid medications.
6. Absence of current severe systemic disease (including, but not limited to: coronary artery disease, chronic obstructive pulmonary disease, congestive heart failure, cancer, and chronic renal disease).
7. Agrees not to undergo any additional weight loss interventional procedures or liposuction for 12 months following study enrollment.
8. Have not taken any prescription or over the counter weight loss medications OR those that can suppress appetite/induce weight loss for at least 6 months and agrees not to utilize for 12 months following study enrollment (including all stimulant medication).
9. Subjects must be willing to possibly forego any future weight loss procedures (i.e. Vertical Sleeve Gastrectomy) given the unknown long-term effects.

Exclusion Criteria:

1. History of (or intra-operative evidence of) prior bariatric, gastric or esophageal surgery.
2. Esophageal stricture or other anatomy and/or condition that could preclude passage of endoluminal instruments or procedure execution.
3. Moderate gastro-esophageal reflux disease (GERD), defined as symptoms that cause subject severe discomfort, compromise performance of daily activities, and/or condition is not entirely controlled with drug therapy.
4. Large hiatal hernia (>3 cm) by history or as determined by pre-enrollment endoscopy.
5. Pancreatic insufficiency/disease.
6. History of gastroparesis or symptoms that would be suggestive of gastroparesis or generalized dysmotility (e.g. esophago-gastric motility issues and lower esophageal sphincter abnormalities).
7. Pregnancy or plans of pregnancy in the next 12 months.
8. Immunosuppressive medications or systemic steroids (i.e., oral prednisone) within 1 month of Visit 1. Intranasal/inhaled steroids are acceptable.
9. History of inflammatory disease of the GI tract; coagulation disorders; hepatic insufficiency or cirrhosis.
10. Active gastric erosion, lesion, or gastric/duodenal ulcer.
11. History of or current platelet or coagulation dysfunction.
12. History or present use of insulin or insulin derivatives for treatment of diabetes.
13. Type II Diabetes Mellitus (as defined by HgbA1c >6.5%) for greater than 11 years at the time of enrollment.
14. If smoker, plans to quit smoking in the year after enrollment.
15. Portal hypertension and/or varices.
16. Patient has a history of drug or alcohol abuse or positive at screening for drugs of abuse.
17. Present or past history of psychosis, bipolar disease, or obsessive-compulsive disorder after pre-enrollment history and medical /psychological assessment.
18. Beck Depression Inventory (Short) Score ≥ 12 and/or uncontrolled depression after pre-enrollment psychological and medical assessment. 1
19. Non-ambulatory or has significant impairment of mobility (i.e. cannot ambulate for 30 minutes).
20. Known hormonal or genetic cause for obesity including untreated hypothyroidism (TSH >5.0 U/ml).
21. Participating in another clinical study.
22. Subjects with a personal history of allergic/anaphylactic reactions including hypersensitivity to the drugs or materials that will be utilized in the study procedure.
23. Physician's assessment that the subject is not an appropriate candidate. If significant findings for depression and/or suicidal ideation are identified, the psychologist(s) assigned to the study will be contacted and arrangement will be made for immediate intervention according to the Institution's standard procedure.

Ages: 22 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Current patients of Roman Turro, MD at Centro Medico Teknon in Barcelona, Spain and Gontrand Lopez-Nava, MD at Madrid Sanchinarro University Hospital in Madrid, Spain
Sampling Method: Non-Probability Sample
Enrollment: 39 (Actual)
Dates: Start 2018-09-18 (Actual); Primary Completion 2020-02-21 (Actual); Study Completion 2020-02-21 (Actual)

PRIMARY OUTCOMES:
Mean % TBWL at 12 months | 12 months
  What is the Mean % TBWL for all Subjects at 12 months
Percentage of subjects with greater than/equal to 5% TBWL at 12 months | 12 months
  What % of subjects who have greater than/equal to 5% TBWL at 12 months
Incidence of Procedure/device related Adverse Events thru 12 months | 12 months
  Overall incidence of procedure/device related adverse events thru 12 months

SECONDARY OUTCOMES:
Change from baseline in gastric emptying test results at 2 and 6 months | 2 & 6 months
  Gather Info on correlation of gastric emptying testing with weight loss outcome

CONTACTS AND LOCATIONS:
Overall Officials: Roman Turro, MD, Principal Investigator — Centro Medico Teknon; Gontrand Lopez-Nava, MD, Principal Investigator — Madrid Sanchinarro University Hospital; Barham Abu Dayyeh, MD, Principal Investigator — Mayo Clinic
Locations (2):
- Spain (2):
  - Centro Medico Teknon, Barcelona
  - Madrid Sanchinarro University Hospital, Madrid

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lopez Nava G, Arau RT, Asokkumar R, Maselli DB, Rapaka B, Matar R, Bautista I, Espinos Perez JC, Bilbao AM, Jaruvongvanich V, Vargas EJ, Storm AC, Neto MG, Abu Dayyeh BK. Prospective Multicenter Study of the Primary Obesity Surgery Endoluminal (POSE 2.0) Procedure for Treatment of Obesity. Clin Gastroenterol Hepatol. 2023 Jan;21(1):81-89.e4. doi: 10.1016/j.cgh.2022.04.019. Epub 2022 May 6. PMID 35533995